CLINICAL TRIAL: NCT02835053
Title: Frailty and Postoperative Outcomes After Emergency General Surgery
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: DM3
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: General Surgery; Geriatrics; Outcomes Research

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Emergency General Surgery: All patients having emergency general surgery procedures as defined by Scott et al (JAMA Surgery 2016)
  Interventions: Other: Frailty

INTERVENTIONS:
Other: Frailty — Participants will be defined as frail based on the Johns Hopkins ACG Frailty Defining Diagnoses Indicator, which will be applied to available health administrative data in the 3 years preceding index hospital admission. If no frailty defining diagnoses are present participants will be defined as not frail

SUMMARY:
The investigators will examine the association between preoperative frailty and postoperative outcomes and resource utilization after emergency general surgery.

ELIGIBILITY:
Inclusion Criteria:

* All residents of Ontario aged more than 65 years on their surgery date with valid provincial health insurance who have an emergency general surgery procedure (large bowel surgery, small bowel surgery, cholecystectomy, control of hemorrhage from duodenal ulcer, lysis of adhesions, appendectomy, laparotomy)

Exclusion Criteria:

* No valid provincial health insurance

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All adult residents of Ontario with valid provincial health insurance who have an emergency general surgery procedure (large bowel surgery, small bowel surgery, cholecystectomy, control of hemorrhage from duodenal ulcer, lysis of adhesions, appendectomy, laparotomy)
Sampling Method: Non-Probability Sample
Enrollment: 150000 (Actual)
Dates: Start 2002-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Mortality | 365 days (from date of surgery)
  Mortality events will be identified from the registered person's database in Ontario from the date of surgery to 365 days after surgery, at which time participants will be censored

SECONDARY OUTCOMES:
Hospital length of stay | day of surgery to 365 days after surgery
  Number of days in hospital from date of surgery to 365 days after surgery
Intensive care unit admission | from date of surgery to 30 days after surgery
  Presence of a special care unit admission from the Discharge abstract database from the date of surgery to 30 days after surgery
Institutional discharge | Date of surgery to hospital discharge or 365 days after surgery (at which time participants will be censored)
  Discharge disposition to an institution in the discharge abstract database
Costs | day of surgery to 365 days after surgery
  Total costs incurred by the provincial health care system from the day of surgery to 365 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided